CLINICAL TRIAL: NCT03082898
Title: Mobility and Therapeutic Benefits Resulting From Exoskeleton Use in a Clinical Setting (SC140121 Study 1 and 2)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Michael Goldfarb, Professor Of Physical Medicine, Vanderbilt University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SC140121
Record Dates: First submitted 2017-02-22; First posted 2017-03-17 (Actual); Results first posted 2022-02-16 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-01

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- AIS A or B using Indego Exoskeleton (Experimental): Patients with American Spinal Injury Association Injury Scale (AIS) A or B (non- ambulatory) will receive regular dosing of exoskeleton walking.
  Interventions: Device: Indego Exoskeleton
- AIS C or D using Indego Exoskeleton (Experimental): Patients with American Spinal Injury Association Injury Scale (AIS) C or D (Poorly ambulatory) will receive regular dosing of exoskeleton walking.
  Interventions: Device: Indego Exoskeleton

INTERVENTIONS:
Device: Indego Exoskeleton — Regular dosing of Indego Exoskeleton walking.

SUMMARY:
The proposed study is intended to inform the hypotheses that (1) regular dosing of exoskeleton walking will provide health benefits to non-ambulatory and poorly-ambulatory individuals with SCI, including decreased pain and spasticity, improvements in bowel and bladder function, decreased body-mass index (BMI), enhanced well-being; (2) regular dosing of exoskeleton walking will facilitate neurological or functional recovery in some individuals with SCI, particularly those with incomplete injuries; and (3) the level of mobility enabled by a lower limb exoskeleton is commensurate with the walking speeds, distances, and surfaces required for community ambulation.

DETAILED DESCRIPTION:
Study Outline Study 1, as described herein, will assess the three hypotheses, i.e., health benefit, neurological recovery, and mobility benefits, in the context of regular dosing of exoskeleton walking in a clinical setting. These studies will be conducted at three study sites, Vanderbilt University Medical Center in Nashville TN, the James A. Haley Veterans Hospital in Tampa FL, and the Mayo Clinic in Rochester MN. All study sites will conduct an identical study protocol. The study will involve 24 non-ambulatory and poorly-ambulatory individuals with incomplete and complete SCI (i.e., 8 subjects at each site). In this study, "poorly ambulatory" is defined as persons with functional independence measure (FIM) gait score of 2 to 6 who may be able to walk short distances with or without braces and stability aid, or may be able to walk with assistance of one person, but whose primary means of mobility is a manual or power-operated wheelchair. Of the 24 individuals, half will be individuals with motor-complete injuries (i.e., American Spinal Injury Association Injury Scale, AIS, A or B), and half with motor-incomplete injuries (i.e., AIS C or D). As described subsequently in the Study Procedures section, the study will assess the therapeutic and functional effects of exoskeleton walking over an 8-week period of treatment, where the treatment consists of 3 walking sessions per week, each approximately 1.5 hours in duration for a total of 24 walking sessions. Therapeutic effects will be assessed via a number of measurements recorded primarily at study start, at the 4-week study midpoint, at the 8-week completion of treatment, and in a follow-up session, 8 weeks following the conclusion of treatment.

Study 2 will add 10 channels of functional electrical stimulation (FES )to the Indego exoskeleton , which include the quadriceps, hamstrings, gastrocnemius, and tibialis anterior muscle groups of each leg, in addition to a pair of trunk muscle channels. The nature of stimulation is fully consistent with standard-of-care FES units, although the timing and amplitude of the leg muscle stimulation is adjusted automatically by the exoskeleton, in a manner similar to the automated adjustment of stimulation in FES-aided cycling devices (also a standard intervention).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.
* Size and limb proportions capable of fitting in the exoskeletal device :
* Height between 1.55 m (5 ft, 1 in) and 1.92 m (6 ft, 3 in).
* Femur length between 37.5 cm (15 in) and 43.125 cm (17.25 in).
* Body mass no greater than 114 kg (250 lb).
* Non-ambulatory or poorly-ambulatory. In this study, "non-ambulatory" is defined as a person who cannot walk, or is classified with a Functional Independence Measure (FIM) Gait score 1; "poorly ambulatory" is defined as a person with FIM Gait 2- 6, who may be able to walk short distances with or without braces or stability aid, or may be able to walk with assistance of one person, but whose primary means of mobility is a manual or power-operated wheelchair.
* Sufficient upper extremity strength and coordination to balance using a appropriate stability aids, such as a rolling walker or forearm crutches, during exoskeleton walking.
* For Study 1 Present with SCI and NLI C5 or lower, with AIS A, B, C or D (as per the International Standard for Neurological Classification of SCI, ISNCSCI), who are non-ambulatory or poorly ambulatory.
* For Study 2: Present with SCI AIS classification A or B at neurological injury level (NLI) T4 or below, or with AIS classification C or D at neurological injury level C5 or below.
* Chronic SCI: at least 6 months post-injury, and preferably post-injury more than 1 year.
* Sufficient bone health for walking with full weight-bearing without undue risk of fracture, as determined by each subject's personal medical doctor, and approved by each site's medical supervisor.
* Passive range of motion (PROM) at shoulders, trunk, upper extremities and lower extremities within functional limits for safe gait and use of appropriate assistive device/stability aid.
* Skin intact where interfacing with robotic device.
* MAS for spasticity score 3 or less in lower extremities.
* Resting Blood pressure and heart rate within established guidelines for locomotor training, specifically: At rest: systolic 150 mmHg or less, diastolic 90 mmHg or less, heart rate 105 bpm or less. During exercise: systolic 180 mmHg or less, diastolic 105 mmHg or less, heart rate 145 bpm or less for Study 1.
* Ability to tolerate an upright standing position for 20 min, passive or active, without being lightheaded or having a headache.
* Sufficient responsiveness to FES in the quadriceps, hamstrings, tibialis anterior, and gastrocnemius, as defined by MMT in response to stimulation of 3 or greater on a 5-point MMT scale. Note that this is specifically for Study 2, but is included in Study 1 in order to economize study resources regarding enrollment, training, and assessment, as previously discussed.
* Access to a wireless internet connection. Note that is required only for Study 3, but is included in Study 1 in order to economize study resources regarding enrollment, training and assessment, as previously discussed.

Exclusion Criteria:

* Heterotopic ossification that, in the opinion of the site medical supervisor, would place the subject at undue risk for fracture.
* Inability to follow instructions.
* Colostomy bag.
* Women who are pregnant or attempting to become pregnant during the course of the study. Note that a pregnancy test will be required and must be negative for all women prior to enrolling in the study, and will be additionally required and must be negative every four weeks during the course of the study protocol.
* Any disease, concomitant injury, or condition that interferes with the performance or interpretation of the protocol- specified assessments.
* Insufficient availability to complete study.
* Any other issue which, in the opinion of the investigators or medical supervisor, make the subject unsuitable for study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-11-15 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Goldfarb, MD, Principal Investigator — Vanderbilt University
Locations (3):
- United States (3):
  - Tampa VA, Tampa, Florida
  - Mayo Clinic, Rochester, Minnesota
  - Vanderbilt, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 41 participants enrolled, 2 were scheduled to start assessments in Tampa, but the study was cancelled due to COVID and not restarted at the Tampa site.
Period: Overall Study
Arm/Group | AIS A or B Using Indego Exoskeleton | AIS C or D Using Indego Exoskeleton
Started | 27 | 12
Completed | 24 | 11
Not Completed | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AIS A or B Using Indego Exoskeleton | AIS C or D Using Indego Exoskeleton | Total
Number analyzed (Participants) | 24 | 11 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 11 | 35
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 19 | 8 | 27
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Time Required to Walk 10 Meters in Seconds as Measured by the Ten Meter Walk Test (10MWT)
Description: Measure of mobility (specifically gait speed) while wearing exoskeleton
Time Frame: Session 11 (Week 5), Session 16 (Week 6), Session 24 (Week 9), and Session 29 (Week 11)
Population: * One participant in the 'AIS A or B using Indego Exoskeleton' group missed the clinic visit for session 24 and we were unable to capture the 10MWT from this participant.
  * One participant in the 'AIS C or D using Indego Exoskeleton' group missed the clinic visit for session 11 and we were unable to capture the 10MWT from this participant.
Measure: Median (Inter-Quartile Range); unit: Seconds
Arm/Group | AIS A or B Using Indego Exoskeleton | AIS C or D Using Indego Exoskeleton
Number analyzed (Participants) | 24 | 11
Seconds
  10MWT at Session 11 (Week 5): number analyzed (Participants) | 24 | 10
  10MWT at Session 11 (Week 5) | 38.3 [33.7 to 49.1] | 28.0 [24.7 to 35.8]
  10MWT at Session 16 (Week 6) | 37.2 [31.4 to 43.0] | 27.9 [25.0 to 33.4]
  10MWT at Session 24 (Week 9): number analyzed (Participants) | 23 | 11
  10MWT at Session 24 (Week 9) | 34.3 [30.3 to 44.3] | 28.6 [26.9 to 32.3]
  10MWT at Session 29 (Week 11) | 32.6 [28.5 to 36.0] | 28.9 [27.5 to 31.7]

2. Primary Outcome: The Total Distance Walked by the Patient in 6 Minutes as Measured by the Six-Minute Walk Test (6MWT)
Description: Measure of gait speed over six minutes while wearing exoskeleton
Time Frame: Session 16 (Week 6) and Session 29 (Week 11)
Measure: Median (Inter-Quartile Range); unit: Feet
Arm/Group | AIS A or B Using Indego Exoskeleton | AIS C or D Using Indego Exoskeleton
Number analyzed (Participants) | 24 | 11
Feet
  6MWT at Session 16 (Week 6) | 288.9 [223 to 332] | 379 [329 to 470]
  6MWT at Session 29 (Week 11) | 297 [250 to 368] | 390 [341 to 400]

3. Secondary Outcome: Time Required to Independently Sit, Stand, Walk, Turn, and Return to Sitting as Measured by the Timed Up and Go (TUG) Test
Description: Measure of ability to stand, walk, turn, and sit while wearing exoskeleton
Time Frame: Session 15 (Week 6), and Session 28 (Week 10)
Measure: Median (Inter-Quartile Range); unit: Seconds
Arm/Group | AIS A or B Using Indego Exoskeleton | AIS C or D Using Indego Exoskeleton
Number analyzed (Participants) | 24 | 11
Seconds
  TUG test at Session 15 (Week 6) | 87.2 [67 to 108] | 66 [61.6 to 93.1]
  TUG test at Session 28 (Week 10) | 84.3 [61.9 to 98.5] | 61.5 [55.8 to 76.0]

ADVERSE EVENTS:
Time Frame: From date of randomization to the follow-up visit at week 18 (session 31)
Description: Adverse event information was collected for any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Groups:
- AIS A or B Using Indego Exoskeleton: Patients with American Spinal Injury Association Injury Scale (AIS) A or B (non- ambulatory) will receive regular dosing of Indego Exoskeleton walking.
- AIS C or D Using Indego Exoskeleton: Patients with American Spinal Injury Association Injury Scale (AIS) C or D (Poorly ambulatory) will receive regular dosing of Indego Exoskeleton walking.
Arm/Group | AIS A or B Using Indego Exoskeleton | AIS C or D Using Indego Exoskeleton
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/11
Other Adverse Events (participants affected / at risk) | 0/24 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2016-02-04): https://cdn.clinicaltrials.gov/large-docs/98/NCT03082898/Prot_000.pdf
  • Statistical Analysis Plan (2016-02-04): https://cdn.clinicaltrials.gov/large-docs/98/NCT03082898/SAP_001.pdf
  • Informed Consent Form (2016-02-04): https://cdn.clinicaltrials.gov/large-docs/98/NCT03082898/ICF_002.pdf